CLINICAL TRIAL: NCT02153268
Title: Phase I/II Open Label FIH Single Center Clinical Study Aimed to Evaluate the Safety and the Efficacy of BonoFill in Reconstructing the Bone.
Brief Title: Filling Bone Defects/Voids With Autologous BonoFill For Maxillofacial Bone Regeneration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: BonusBio Group Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-BNS-02
Record Dates: First submitted 2014-04-20; First posted 2014-06-03 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Bone Void in the Maxillofacial Area
Keywords: Safety; efficacy; BonoFill; bone filler; autologous adipose tissue derived cells (HATDCs); Bone augmentation; sinus augmentation; Bone grafting after removal of cysts from jaws

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- single arm, Liposuction, BonoFill Transplantation (Experimental): * Liposuction - will be performed on Visit 2 for all eligible subjects
  * BonoFill Transplantation - will be performed on Visit 6 for all eligible subjects
  Interventions: Procedure: Single Arm - Liposuction procedure and BonoFill transplantation will be done for all subjects on study

INTERVENTIONS:
Procedure: Single Arm - Liposuction procedure and BonoFill transplantation will be done for all subjects on study — Liposuction - will be performed on Visit 2, BonoFill will be based on subject's autologous Human Adipose Tissue Derived Cells (HATDCs).
  BonoFill Transplantation will be performed on Visit 6. BonoFill will be administrated to the subject in a single session at one tested cell dose.
  Other Names: BonoFill is an Biological, cell therapy Product that complies with the definition of Somatic Cell Therapies; BonoFill is an autologous Human Adipose Tissue Derived Cells (HATDCs) based product, combined with OraGraft® mineral particles.

SUMMARY:
Phase I/II open label first in human single center clinical study, is to evaluate the safety and the efficacy of BonoFill as bone filler containing the patient own (autologous) adipose tissue derived cells (HATDCs) in reconstructing the Bone Void in the maxillofacial area approximately 6 month follow up after implantation in the following two clinical indications:

1. Bone augmentation (e.g. sinus augmentation)
2. Bone grafting after removal of cysts from jaws

DETAILED DESCRIPTION:
Primary endpoint: The implantation of BonoFill to the maxillary or mandible defect/void is safe under the following conditions: No chronic bone infection (Osteomyelitis); no significant changes in complete blood count (CBC) and in general health.

Secondary endpoint: The implantation of BonoFill to the maxillary or mandible void is efficient under the following conditions: Following BonoFill implantation, the bone regeneration in the operated site was significantly accelerated. Also, the bone defects/voids were filled with a significant amount of bone tissue.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria defining the eligible subjects are divided to two groups according clinical indications:

Sinus augmentation

* Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs physical examination and safety lab tests
* Subjects that have a rehabilitation dentist and rehabilitation program
* Up to dated panoramic X-Ray.
* Subjects who provided written informed consent to participate in the study, able to understand study procedure and agree for follow up procedures
* Healthy conditions of Maxillary Sinuses and Oral Mucosa.
* Sub-antral bone at least 4 mm as measured on CBCT/CT.
* Have a good oral hygiene condition as per investigator discretion.

Bone grafting after removal of cysts from jaws

* Healthy subject.
* Subjects that have a rehabilitation dental treatment.
* Limited to cysts diagnosed as: radicular cysts, residual cysts, congenital cysts, developmental and acquired cysts.
* Subjects referred to oral & maxillofacial Dpt for removal of cysts after diagnosis of the cyst type.
* Healthy bone determined by X-ray.
* Have a good oral hygiene condition.
* Subject that does not participate in other clinical study.
* Subject able to read and understand and sign the informed consent

Exclusion Criteria:

* Subjects with recorded medical history diseases as: diabetes mellitus, heart diseases, renal failure, osteoporosis.
* Subject treated with systemic steroid treatment
* Subjects with known autoimmune diseases, such as: Addison's disease Celiac disease - sprue (gluten-sensitive enteropathy), Dermatomyositis Graves disease, Hashimoto's thyroiditis, Multiple sclerosis, Myasthenia gravis Pernicious anemia, Reactive arthritis, Rheumatoid arthritis, Sjogren syndrome Systemic lupus erythematosus, Type I diabetes.
* Subjects that have Vitiligo and/or known scar healing problems (keloid formation).
* Subjects treated with anticoagulation medication (such as Coumadin, Plavix and other similar medications)
* Subjects treated with Oral Bisphosphonate drugs (such as Fosalan and other similar medications)
* Subjects with a history of Chemotherapy or Radiotherapy treatment
* In case of sinus augmentation - Unhealthy conditions of Maxillary Sinuses.
* Subjects with current active infection or illness
* Subjects participating in another clinical trial 30 days prior to and during the study period
* Pregnant or lactating woman. Pregnancy will be verified by urine test during screening
* Known history of any significant medical disorder, which in the investigator's judgment contraindicates the subject's participation
* Subjects with any known allergy for anesthesia
* Positive serology for either HIV, hepatitis B or hepatitis C
* Abnormal clinically significant as per investigator's judgment laboratory test and exams findings

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
BonoFill is safe | approximately 6 month follow up after implantation
  The implantation of BonoFill to the maxillary or mandible defect/void is safe under the following conditions: No chronic bone infection (Osteomyelitis); no significant changes in complete blood count (CBC) and in general health.

SECONDARY OUTCOMES:
BonoFill is efficient | approximately 6 month follow up after implantation
  The implantation of BonoFill to the maxillary or mandible void is efficient under the following conditions: Following BonoFill implantation, the bone regeneration in the operated site was significantly accelerated. Also, the bone defects/voids were filled with a significant amount of bone tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Stolero, Dr, Principal Investigator — MY
Locations (1):
- Dr. Ephraim Zur Dental Clinic, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: No